CLINICAL TRIAL: NCT00652054
Title: An Open-Label, Non-Randomized, Multicenter, Two-Stage, Phase 2 Study of S-1 as 2nd Line Therapy for Patients With Metastatic Pancreatic Cancer Who Have Previously Received 1st Line Treatment With a Gemcitabine Regimen
Brief Title: Phase 2 Study of S-1 as 2nd Line Therapy in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Fabio Benedetti, M.D., Chief Medical Officer, Taiho Pharma USA, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1201; NCT00227604 (obsolete NCT alias)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All patients will receive S-1 orally at a dose of 30 mg/m2 twice daily (BID) for 14 days followed by a 1-week recovery period, repeated every 3 weeks.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — All patients will receive S-1 orally at a dose of 30 mg/m2 twice daily (BID) for 14 days followed by a 1-week recovery period, repeated every 3 weeks. The trial will proceed to the second stage only if sufficient efficacy is demonstrated in Stage 1.

SUMMARY:
The purpose of this study is to determine whether S-1 is effective as 2nd line therapy in slowing tumor activity in patients with metastatic pancreatic cancer who have previously received 1st line treatment with a gemcitabine regimen. The study is also looking at the safety of S-1.

DETAILED DESCRIPTION:
Metastatic pancreatic cancer is relatively unresponsive to chemotherapy. This is true for the nucleoside analogue gemcitabine, with a response rate of approximately 10%, as well as for 5-fluorouracil (5-FU). Even when gemcitabine is combined with other chemotherapeutic drugs or biological agents, the overall tumor response rate remains basically unchanged. S-1 is a new generation oral fluoropyrimidine that combines Tegafur (5-fluoro-1-(tetrahydro-2-furanyl)-2,4(1H,3H)-pyrimidinedione [FT]), an oral prodrug of 5-FU, with two modulators, Gimeracil (5-chloro-2,4-dihydroxypyridine [CDHP]), which inhibits 5-FU degradation by dihydropyrimidine dehydrogenase (DPD) inhibition, and Oteracil potassium (Oxo), which inhibits 5-FU phosphorylation in the digestive tract. This combination of 3 compounds is designed to achieve enhanced antitumor activity while decreasing gastrointestinal toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 1. Has provided written informed consent. 2. Has histologically or cytologically confirmed locally advanced, unresectable or metastatic adenocarcinoma of the pancreas not amenable to curative radiotherapy or surgery.

  3. Has measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (ie, lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm using spiral computed tomography [CT] scan).

  4. Is able to take medications orally. 5. Is 18 years of age or older. 6. Has a Karnofsky Performance Status (KPS) ≥ 70% (see Appendix A). 7. Has a life expectancy of ≥ 12 weeks. 8. Has adequate organ function as defined by the following criteria:
  1. Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times the upper limit of normal (ULN). If liver function abnormalities are due to underlying liver metastasis, then AST (SGOT) and ALT (SGPT) may be ≤ 5 times ULN.
  2. Total serum bilirubin ≤ 3.0 times ULN (if due to underlying liver metastasis, then total bilirubin may be ≤ 5 times ULN).
  3. Absolute granulocyte count ≥ 1,500/mm3 (ie, ≥ 1.5 x 109/L by International Units [IU]).
  4. Platelet count ≥ 100,000/mm3 (IU: ≥ 100 x 109/L).
  5. Hemoglobin value ≥ 9.0 g/dL.
  6. Calculated creatinine clearance ≥ 60 mL/min (based on serum creatinine) (Cockcroft-Gault85 formula) 9. Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

     Exclusion Criteria:
* 1. Has had treatment with any of the following within the specified time frame prior to study drug administration:

  1. Any prior anticancer chemotherapy.
  2. Radiation therapy to a target lesion unless there was evidence of PD after radiotherapy (and this target lesion must not be the only site of measurable disease).
  3. Any radiotherapy within the previous 3 weeks.
  4. Any investigational agent received either concurrently or within the last 30 days.
  5. Current enrollment in another clinical study with an investigational agent. Patients participating in surveys or observational studies are eligible to participate in this study.

     2. Major surgery within the previous 3 weeks. 3. Symptomatic brain metastasis not controlled by corticosteroids. 4. Leptomeningeal metastasis. 5. Previous or concurrent malignancy other than pancreatic cancer except adequately treated carcinoma in-situ of the cervix or non-melanoma skin cancer. 6. Uncontrolled ascites requiring drainage at least twice a week. 7. Other serious illness or medical condition(s) including, but not limited to, the following:

  <!-- -->

  1. Uncontrolled congestive heart failure (New York Heart Association [NYHA] Class III or IV), angina pectoris, arrhythmias, or hypertension.
  2. Active infection.
  3. Known (at time of entry) gastrointestinal disorder, including malabsorption, chronic nausea, vomiting, or diarrhea, present to the extent that it might interfere with oral intake and absorption of study medication.
  4. Poorly controlled diabetes mellitus.
  5. Psychiatric disorder that may interfere with consent and/or protocol compliance.
  6. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
  7. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.

     8. Is receiving a concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1:

  <!-- -->

  1. Sorivudine, uracil, cimetidine, folinic acid, and dipyridamole (may enhance S-1 activity).
  2. Allopurinol (may diminish S-1 activity).
  3. Phenytoin (S-1 may enhance phenytoin activity).
  4. Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 and flucytosine activity).

     9. Is a pregnant or lactating female. 10. Has known sensitivity to 5-FU. 11. Is a patient with reproductive potential who refuses to use an adequate means of contraception (including male patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Overall tumor response rate (ORR - the proportion of patients with objective evidence of PR or CR) | Each cycle will last 21 days (14 days treatment, 7 days recovery) for 6 mos. Tumor assessmentswill be obtained at baseline) and at the end of every even cycle.

SECONDARY OUTCOMES:
To evaluate the duration of response (DR), progress-free survival (PFS), and survival rate | Each cycle will last 21 days (14 days treatment, 7 days recovery for 6 mos. Pts will be followed for survival status every 2 months following PD for up to 6 mos.
To investigate the effect of S-1 on Karnofsky Performance Status (KPS), weight, and analgesic consumption | KPS and wt measured at baseline; w/in 24 hrs pr study drug on Day 1 of each cycle after Cycle 1; end of study treatment. Info on analgesics gathered at least 7 days prior to Day 1 of Cycle 1 and continuing through end of treatment.
To evaluate CA19-9 decline | Each cycle will last 21 days (14 days treatment, 7 days recovery) for 6 mos. CA19-9 levels will be collected at basleine, Day 1 of each cycle, and at the end of treatment.
To evaluate the safety profile of S-1 | AEs will be reported from the time a patient signs informed consent through the period of patient follow-up Blood/urine will be collected at baseline; Days 8&15; w/in 24 hrs of study drug on Day 1 of each cycle after Cycle 1; at end of study treatment.
To investigate the relationship of S-1 plasma levels (components and metabolites) with safety and efficacy parameters | Each cycle will last 21 days (14 days treatment, 7 days recovery) for 6 mos. Blood samples to be obtained 1.5 ± 0.5 h, 5 ± 1 h, 7 ± 1 h postdose on Day 1 of Cycle 1 only.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Benedetti, MD, Study Director — Taiho Oncology, Inc.